CLINICAL TRIAL: NCT04961398
Title: Evaluation of Heidelberg Engineering SPECTRALIS OCT Signal to Noise Ratio Effect on Parameter Measurements
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: S-2021-1
Record Dates: First submitted 2021-06-17; First posted 2021-07-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Normal Eyes

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- OCT speed 85 KHz: predicate speed
  Interventions: Device: OCT imaging
- OCT speed 125 KHz: investigational speed
  Interventions: Device: OCT imaging
- OCT speed 20 KHz: investigational speed
  Interventions: Device: OCT imaging

INTERVENTIONS:
Device: OCT imaging — OCT imaging on Normal Eyes without any filter and with various ND filters as per protocol

SUMMARY:
Evaluation of effect of various OCT scan speeds and filters on parameter measurements.

DETAILED DESCRIPTION:
The objectives of this study are to

1. Directly compare parameter measurements generated on scans acquired at different speed modes with various levels of signal-to-noise ratio (SNR).
2. Evaluate the effects of SNR, as determined by the device's Q score, on parameters derived from segmentation results, i.e., thickness of peripapillary retinal nerve fiber layer on circle scans (pRNFL), minimum rim width of optical nerve head (MRW), and macular layer thicknesses (Retina, GCL, IPL).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
2. Age ≥ 22
3. Both eyes with an age-appropriate normal appearing OCT as determined by an investigator

Exclusion Criteria:

1. Subjects unable to read or write
2. Subjects with ocular media not sufficiently clear to obtain acceptable study-related imaging as determined by OCT imaging (without neutral optical density filter)
3. Subjects who cannot tolerate the imaging procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with healthy eyes
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Macular layer thicknesses | during the intervention
  ETDRS grid (9 sectors)
Bruch's Membrane Opening (BMO)-Minimum Rim Width (MRW) | during the intervention
  Classification chart (6 sectors)
Peripapillary Retinal Nerve Fiber Layer Thickness (RNFLT) | during the intervention
  Classification chart (6 sectors)

SECONDARY OUTCOMES:
Adverse Events | through study completion, an average of one day
  All AEs

CONTACTS AND LOCATIONS:
Overall Officials: Valerie M Leung, BOptom BS, Principal Investigator — Heidelberg Engineering, Inc.
Locations (1):
- Heidelberg Engineering, Inc., Franklin, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No